CLINICAL TRIAL: NCT04196270
Title: The Minimal Effective Volume (MEV90) of Ropivacaine 0.75% for Ultrasound-guided Transmuscular Quadratus Lumborum Block for Unilateral Percutaneous Nephrolitotomy: a Study Protocol for a Dose Finding Trial
Brief Title: The Minimal Effective Volume (MEV90) of Ropivacaine 0.75% for Ultrasound-guided Transmuscular Quadratus Lumborum Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Clinical Trials Zealand
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: dose finding study
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: The biased coin up-and-down sequential design (BCD) should be considered for direct determination of higher quantiles (ED90 and ED95) which provide useful clinical knowledge. The BCD was developed in the field of pharmacology and toxicology and was formulated by Durham et al. in 1997. In the BCD, volume assignment is carried out in a sequential and interactive method, which avoids that patients are randomized to doses with toxicity risk and seeks to concentrate treatments around the suitable doses.
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ropivacaine (Experimental): This double-blind dose-finding trial is based on a biased coin up-and-down sequential design, where the volume of local anesthetic administered to each patient depends on the response from the previous one. The TQL block is performed preoperatively, and the first patient recruited receives 20 mL of ropivacaine 0.75%. In case of block failure, the next patient will receive a higher volume (defined as the previous volume with an increment of 2 mL). Given a successful block for the first patient, the next patient will be randomized to either a lower volume (defined as the previous volume with a reduction of 2 mL) or the same volume as the previous patient. The respective probabilities being b=0.11 for a reduced volume and 1-b=0.89 for the same volume. Block success is defined as patient reported numeric rated scale (NRS) pain (NRS value ≤ 3 (0-10/10)), 30 minutes after arrival in the post anesthesia care unit (PACU).
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — In a dose finding study the total volume of ropivacaine changes according to the biased coin up-and-down sequential design
  Other Names: Sequential design

SUMMARY:
This double-blind dose-finding trial is based on a biased coin up-and-down sequential design, where the volume of local anesthetic administered to each patient depends on the response from the previous one. The TQL block is performed preoperatively, and the first patient recruited receives 20 mL of ropivacaine 0.75%. In case of block failure, the next patient will receive a higher volume (defined as the previous volume with an increment of 2 mL). Given a successful block for the first patient, the next patient will be randomized to either a lower volume (defined as the previous volume with a reduction of 2 mL) or the same volume as the previous patient. The respective probabilities being b=0.11 for a reduced volume and 1-b=0.89 for the same volume. Block success is defined as patient reported numeric rated scale (NRS) pain (NRS value ≤ 3 (0-10/10)), 30 minutes after arrival in the post anesthesia care unit (PACU). The NRS pain value is our primary and only outcome in the evaluation of the block. A minimum of 25 eligible patients are needed to achieve precise estimation of MEV90 with narrow 95% confidence intervals derived by bootstrapping. Following inclusion of 25 patients early termination is considered when interim analysis shows sufficiently stabilization of MEV90 estimate. The final sample size is not known a priori, but a maximum of 40 patients will be enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the trail must comply with all of the following requirements to be included:

  * Scheduled for elective PNL surgery in general anesthesia with propofol and remifentanil
  * Age > 18 years at the date of inclusion
  * Have received thorough information, oral and written, and signed the "informed consent" form on participation in the trail
  * ASA score 1-3

Exclusion Criteria:

* Inability to speak and understand Danish
* Allergy to local anesthetics or opioids
* Daily intake of opioids (evaluated by the investigators)
* Drug and/or substance abuse
* Local infection at the site of injection or systemic infection
* Difficult visualization of muscular and fascial structures necessary for successful block administration
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-05 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Numeric rated scale | 30 minutes after arrival in the post anesthesia care unit
  Pain score from numeric rated scale 0-10/10 Pain score, numeric rated scale 0-10/10. 0=no pain, 10=maximum pain

IPD SHARING:
Plan to Share IPD: No